CLINICAL TRIAL: NCT06057064
Title: A Phase II Randomized, Double-blind Study to Evaluate the Safety, Neutralizing Activity and Efficacy of AZD3152 for Pre-exposure Prophylaxis of COVID-19 in Participants Having an Increased Risk for Inadequate Response to Active Immunization (NOVELLA)
Brief Title: Study Will Assess the Safety, Neutralizing Activity and Efficacy of AZD3152 in Adults With Conditions Increasing Risk of Inadequate Protective Immune Response After Vaccination and Thus Are at High Risk of Developing Severe COVID-19
Acronym: NOVELLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZ-RU-00002
Record Dates: First submitted 2023-09-26; First posted 2023-09-28 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: COVID-19, SARS-CoV-2
Keywords: Pre-exposure Prophylaxis of COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a Phase II Randomized, Double-blind Study to Evaluate the Safety, Neutralizing Activity and Efficacy of AZD3152 for Pre-exposure Prophylaxis of COVID-19 in adult participants. Approximately 116 participants in Russia will be randomized at up to 10 study sites in a ratio of 3:1 to either AZD3152 or placebo administered IM.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of Placebo IM (0.9% sodium chloride)
  Interventions: Biological: Biological: Placebo
- AZD3152 (Experimental): Single dose of 300 mg IM
  Interventions: Biological: Biological: AZD3152

INTERVENTIONS:
Biological: Biological: AZD3152 — 300 mg single dose of AZD3152 IM
  Arms: AZD3152
Biological: Biological: Placebo — Single dose of Placebo IM (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
AZD3152, a single mAb, is being developed to have broad neutralizing activity across known SARS-CoV-2 variants of concern for pre-exposure prophylaxis of COVID-19.

The aim of the Phase II study is to evaluate the safety, neutralizing activity and efficacy of AZD3152 for pre exposure prophylaxis of COVID-19

DETAILED DESCRIPTION:
Phase II study to assess the safety, neutralizing activity and efficacy of one dose of AZD3152 compared with one dose of placebo in adults with immunocompromised conditions, including comorbidities contributing to weakened immunity, thereby increasing the risk of COVID-19 progression up to severe grade.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or older at the time of signing the informed consent.
* Weight ≥ 45 kg at Visit 1.
* Participants must satisfy at least 1 of the following risk factors at enrollment:

  1. Obese, ie, BMI ≥ 30
  2. Congestive heart failure
  3. Chronic obstructive pulmonary disease
  4. Chronic kidney disease
  5. Intolerant of vaccine
  6. Immunocompromised state (one of the following risk factors ):

     1. Have cancer
     2. Have solid organ transplant or a hematopoietic stem cell transplant
     3. Are actively taking immunosuppressive medicines
     4. Received chimeric antigen receptor T-cell therapy
     5. Within 1 year of receiving B-cell depleting therapies
     6. Have a moderate or severe primary immunodeficiency
* Medically stable
* WOCBP must not be pregnant or lactating and must use a highly effective method of contraception

Exclusion Criteria:

* Known hypersensitivity to any component of the study intervention
* Previous hypersensitivity or severe adverse reaction following administration of a mAb
* Acute or febrile infection prior to dosing
* Has HIV infection
* Receipt of any convalescent COVID-19 plasma treatment, mAb against SARS-CoV-2 , COVID-19 vaccine within 6 months
* COVID-19 antiviral prophylaxis within at least 2 weeks
* COVID-19 case within 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. All the data will be provided in blinded manner until final unblinded data analysis will be completed. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=AZ-RU-00002&attachmentIdentifier=6f37b4ef-51bd-4c91-8219-cdb0a98770d3&fileName=AZ-RU-00002_CSP_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=AZ-RU-00002&attachmentIdentifier=a16b9586-8ea9-4bce-bda0-d1d777305a9e&fileName=AZ-RU-00002_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=AZ-RU-00002&attachmentIdentifier=14cb7005-83a5-4842-aade-23ba6c51f461&fileName=AZ-RU-00002_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: [Not Specified]
Pre-assignment Details: [Not Specified]
Groups:
- AZD3152: AZD3152 300 mg
- Placebo: Saline Placebo
Period: Overall Study
Arm/Group | AZD3152 | Placebo
Started | 87 | 29
Completed (111) | 83 | 28
Not Completed | 4 | 1
Not completed — Death | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD3152 | Placebo | Total
Number analyzed (Participants) | 87 | 29 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (12.61) | 58.2 (11.78) | 56.2 (12.41)
Age, Customized [Number; unit: Participants]
  >= 18 to <60 years | 52 | 15 | 67
  >=60 years | 35 | 14 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 17 | 61
  Male | 43 | 12 | 55
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 83 | 28 | 111
  Missing | 4 | 1 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 86 | 29 | 115
  Asian | 1 | 0 | 1
  Other | 0 | 0 | 0
  Not Reported | 0 | 0 | 0
Previous COVID-19 vaccinations [Number; unit: Participants] | 56 | 13 | 69
SARS-CoV-2 status at baseline [Count of Participants; unit: Participants]
  Negative | 87 | 29 | 116
  Positive | 0 | 0 | 0
  Missing | 0 | 0 | 0
Any COVID-19 comorbidities at baseline [Count of Participants; unit: Participants]
  Yes | 87 | 29 | 116
  Missing | 0 | 0 | 0
Any high risk for severe COVID-19 [Count of Participants; unit: Participants]
  Yes | 87 | 29 | 116
  Missing | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 171.0 (9.39) | 170.7 (8.80) | 170.9 (9.21)
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (6.08) | 27.8 (5.30) | 28.5 (5.89)

OUTCOME MEASURES:

1. Primary Outcome: The Number and Proportion of Subjects With AEs, SAEs, MAAEs, AESIs.
Description: The safety profile will be evaluated using vital signs, laboratory data, electrocardiograms (ECGs), and adverse event data
Time Frame: up to Day 181
Population: Safety analysis population
Measure: Count of Participants; unit: Participants
Arm/Group | AZD3152 | Placebo
Number analyzed (Participants) | 87 | 29
Participants
  Adverse Events | 45 | 17
  Serious Adverse Events | 5 | 2
  Medically Attended Adverse Events | 14 | 7
  Adverse Events of Special Interest | 0 | 0

2. Secondary Outcome: Geometric Mean Titer (GMT) of nAbs Against SARS-CoV-2 Emerging Dominant Variant(s)
Description: GMT of nAbs against SARS-CoV-2 emerging dominant variant(s) circulating during the course of the study (measured in RU local laboratory)
Time Frame: up to Day 181
Population: SARS-CoV-2 nAb Set
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | AZD3152 | Placebo
Number analyzed (Participants) | 87 | 29
Titer
  Baseline GMT | 12.0 (3.22) | 9.8 (2.50)
  Visit 2. Day 8 GMT: number analyzed (Participants) | 87 | 28
  Visit 2. Day 8 GMT | 67.7 (2.02) | 11.3 (2.76)
  Visit 3. Day 15 GMT: number analyzed (Participants) | 86 | 29
  Visit 3. Day 15 GMT | 70.9 (1.96) | 12.1 (2.89)
  Visit 4. Day 29 GMT: number analyzed (Participants) | 76 | 27
  Visit 4. Day 29 GMT | 64.3 (2.05) | 12.6 (2.67)
  Visit 5. Day 91 GMT: number analyzed (Participants) | 67 | 22
  Visit 5. Day 91 GMT | 37.6 (2.24) | 9.1 (2.25)
  Visit 6. Day 181 GMT: number analyzed (Participants) | 61 | 19
  Visit 6. Day 181 GMT | 22.4 (2.71) | 13.4 (2.76)

3. Secondary Outcome: Geometric Mean Fold Rise (GMFRs) of nAb Titers Against SARS-CoV-2 Emerging Dominant Variant(s)
Description: GMFR (from baseline) of nAb titers against SARS-CoV-2 emerging dominant variant(s) circulating during the course of the study (measured in RU local laboratory)
Time Frame: up to Day 181
Population: SARS-CoV-2 nAb Set
Measure: Geometric Mean (Standard Deviation); unit: fold rise
Arm/Group | AZD3152 | Placebo
Number analyzed (Participants) | 87 | 29
fold rise
  Visit 2. Day 8 GMFRs: number analyzed (Participants) | 87 | 28
  Visit 2. Day 8 GMFRs | 5.63 (2.663) | 1.16 (1.941)
  Visit 3. Day 15 GMFRs: number analyzed (Participants) | 86 | 29
  Visit 3. Day 15 GMFRs | 5.84 (2.491) | 1.24 (2.247)
  Visit 4. Day 29 GMFRs: number analyzed (Participants) | 76 | 27
  Visit 4. Day 29 GMFRs | 4.71 (2.295) | 1.33 (2.014)
  Visit 5. Day 91 GMFRs: number analyzed (Participants) | 67 | 22
  Visit 5. Day 91 GMFRs | 2.81 (2.653) | 1.10 (1.986)
  Visit 6. Day 181 GMFRs: number analyzed (Participants) | 61 | 19
  Visit 6. Day 181 GMFRs | 1.71 (2.565) | 1.55 (2.462)

4. Secondary Outcome: Incidence of a Post-treatment Symptomatic COVID-19 Case
Description: Incidence of a post-treatment symptomatic COVID-19 case (negative RT-PCR at baseline to positive RT-PCR or positive antigen test at any time up to 6 months AND symptoms specified in the modified WHO definition of symptomatic COVID-19).
Time Frame: up to Day 181
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | AZD3152 | Placebo
Number analyzed (Participants) | 87 | 29
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: AEs, MAAE, AESI will be collected from the time of study intervention administration throughout the study, up to and including the last visit, an average of 6 months. SAEs will be recorded from the time of signing of the ICF throughout the study, up to and including the last visit, an average of 6 months.
Arm/Group | AZD3152 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/87 | 0/29
Serious Adverse Events (participants affected / at risk) | 5/87 | 2/29
Other Adverse Events (participants affected / at risk) | 45/87 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AZD3152 (N=87) | Placebo (N=29)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Necrotising ulcerative gingivostomatitis (Infections and infestations) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1/1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD3152 (N=87) | Placebo (N=29)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (2)
Chest pain (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 9 (10) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (3)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Acute sinusitis (Infections and infestations) | 3 (4) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (3)
Oral herpes (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Necrotising ulcerative gingivostomatitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otosalpingitis (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic cystadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Brachiocephalic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT06057064/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT06057064/SAP_001.pdf